CLINICAL TRIAL: NCT03322579
Title: Balloon Dilation of the Eustachian Tube, a Lower Pressure Challenge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0034-17
Record Dates: First submitted 2017-03-28; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Intervention Model Description: Unilateral or bilateral balloon catheter dilation will be performed on patients with eustachian tube dysfunction
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with Eustachian tube dysfunction (Experimental)
  Interventions: Device: Balloon dilatation Eustachian tuboplasty

INTERVENTIONS:
Device: Balloon dilatation Eustachian tuboplasty — Eustachian tuboplasty by balloon dilation involves the recanalization of the cartilaginous portion of the ET via the nasopharynx with a balloon catheter. This catheter is inflated to multiple atmospheres of pressure for a short amount of time and then removed.

SUMMARY:
Balloon dilatation Eustachian tuboplasty has recently become a promising procedure for the treatment of refractory dilatory dysfunction of the Eustachian tube.

Eustachian tube (ET) comprises an osseous intratemporal portion and a cartilaginous nasopharyngeal portion. It functions in pressure equalization, middle ear protection and clearance. Eustachian tube function can be adversely affected by viral and bacterial infections, adenoid disease, craniofacial anomalies, neoplasm, genetic predisposition, sinonasal disease and gastroesophageal reflux, leading to Eustachian tube dysfunction. Eustachian tuboplasty by balloon dilation involves the recanalization of the cartilaginous portion of the ET via the nasopharynx with a balloon catheter. This catheter is inflated to multiple atmospheres of pressure for a short amount of time and then removed.

The surgical technique, the optimal balloon diameter, pressure or duration of inflation are variable in the literature.

Even though the current data shows promising results and a potential benefit of this procedure, further evaluation is still needed in order to establish a higher level of evidence of efficacy and safety.

DETAILED DESCRIPTION:
Balloon dilatation Eustachian tuboplasty has recently become a promising procedure for the treatment of refractory dilatory dysfunction of the Eustachian tube.

Eustachian tube (ET) comprises an osseous intratemporal portion and a cartilaginous nasopharyngeal portion. It functions in pressure equalization, middle ear protection and clearance. Eustachian tube function can be adversely affected by viral and bacterial infections, adenoid disease, craniofacial anomalies, neoplasm, genetic predisposition, sinonasal disease and gastroesophageal reflux, leading to Eustachian tube dysfunction.

it is now well known that the site of pathology is usually in the cartilaginous portion and not within the osseus portion.

Chronic dilatory dysfunction of the Eustachian tube is estimated to be 1% of the adult population. Current medical and surgical treatment options for this pathophysiological disorder is still unsatisfactory, including nasal decongestants, topical and systematic corticosteroids, antihistamines and multiple insertions of ventilation tubes leading to complications.

ET dysfunction can lead to impaired quality of life due to persistent sensation of ear fullness, ear pain and inability to tolerate air travel, diving or other activities. With time, Eustachian tube dysfunction, if left untreated can lead to complications such as conductive hearing loss and cholesteatoma formation. Recently, numerous researches have investigated the role of balloon tuboplasty. This procedure aims to ventilate and drain the middle ear by improving the physiological function of the eustachian tube and treating chronic refractory eustachian tube dysfunction.

Eustachian tuboplasty by balloon dilation involves the recanalization of the cartilaginous portion of the ET via the nasopharynx with a balloon catheter. This catheter is inflated to multiple atmospheres of pressure for a short amount of time and then removed.

The surgical technique, the optimal balloon diameter, pressure or duration of inflation are variable in the literature.

Both cadaveric and clinical studies where done. Cadaveric studies revealed no evidence of fractures to the cartilaginous or bony lumen, and no damage to the internal carotid artery. Several clinical studies and many others that confirm the safety of eustachian tube balloon dilation and consider it as a potential solution for chronic eustachian tube dysfunction. A systematic review preformed in 2014 showed no adverse outcomes in 103 patients who had undergone balloon dilation of the Eustachian tube. Another more recent systematic review in 2016 that included nine prospective studies, describing 713 eustachian tube balloon dilations in 474 patients confirm the safety of eustachian tube balloon dilation.

In September 2016 the ACCLARENT AERA™ Eustachian Tube Balloon Dilation System, has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of Eustachian Tube Dysfunction (ETD) and was permitted for marketing.

Even though the current data shows promising results and a potential benefit of this procedure, further evaluation is still needed in order to establish a higher level of evidence of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (over 18 years) with a diagnosis of Eustachian tube dysfunction based on symptoms and abnor-mal tympanogram.
2. OME and/or TM atelectasis
3. Type B or C tympanograms
4. Inability to inflate middle ears by Valsalva maneuver.
5. Patients performed tympanocentesis and patients underwent tube insertion will be included.

Exclusion Criteria:

1. Children less than 18 years old.
2. Patients with an active infection.
3. Patients with craniofacial abnormalities.
4. Pregnancy?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The change in eustachian tube function | 1,3,6 and 12 month post procedure
  Otoscopy

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607